CLINICAL TRIAL: NCT00096317
Title: The Effect of Ketoconazole on the Pharmacokinetics and Pharmacodynamics of Ixabepilone In Patients With Advanced Cancer
Brief Title: Ixabepilone and Ketoconazole in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000393439; P30CA013330 (NIH); AECM-03099; AECM-CA163402; AECM-NMC-03-10-277C
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — ixabepilone; Ketoconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: ixabepilone
Drug: ketoconazole

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ixabepilone and ketoconazole, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving ixabepilone with ketoconazole may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving ixabepilone together with ketoconazole and to see how well they work in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of ketoconazole on the pharmacokinetics of ixabepilone in patients with advanced solid tumors.

Secondary

* Determine the safety of ixabepilone when administered alone and in combination with ketoconazole in these patients.
* Determine, preliminarily, the antitumor activity of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of ixabepilone.

During course 1, patients receive oral ketoconazole on days 0-5 and ixabepilone IV over 3 hours on day 1. During course 2 and subsequent courses, patients receive only ixabepilone IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of at least 3 patients receive escalating doses of ixabepilone during course 1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose-limiting toxicity. At least 12 patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 3-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor
* Unresponsive to currently available therapy OR no known effective treatment exists
* Measurable or nonmeasurable disease
* Brain metastases allowed, provided the following criteria are met:

  * Completed cranial radiotherapy at least 4 weeks ago
  * Stable or reduced brain metastases by brain imaging*
  * Clinically stable disease AND no steroid therapy within the past 2 weeks (Baseline brain imaging is not required for patients with no signs or symptoms of brain metastasis)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 3 prior chemotherapy regimens
* No other concurrent chemotherapy (standard or investigational)

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to > 25% of major bone-marrow containing areas (e.g., pelvis or lumbar spine)

Surgery

* At least 1 week since prior minor surgery and recovered
* At least 3 weeks since prior major surgery and recovered

Other

* More than 2 weeks since prior drugs that would inhibit or stimulate drug metabolism

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2005-12-05 (Actual); Study Completion 2005-12-05 (Actual)

PRIMARY OUTCOMES:
Effect of ketoconazole on the pharmacokinetics of ixabepilone

SECONDARY OUTCOMES:
Safety of ixabepilone with and without ketoconazole
Antitumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Study Chair — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Result] Goel S, Cohen M, Comezoglu SN, Perrin L, Andre F, Jayabalan D, Iacono L, Comprelli A, Ly VT, Zhang D, Xu C, Humphreys WG, McDaid H, Goldberg G, Horwitz SB, Mani S. The effect of ketoconazole on the pharmacokinetics and pharmacodynamics of ixabepilone: a first in class epothilone B analogue in late-phase clinical development. Clin Cancer Res. 2008 May 1;14(9):2701-9. doi: 10.1158/1078-0432.CCR-07-4151. PMID 18451235